CLINICAL TRIAL: NCT06306560
Title: An Exploratory Clinical Study of Adebrelimab in Combination With Famitinib and Chemotherapy for the Treatment of First-line Extensive Stage Small Cell Lung Cancer
Brief Title: A Study of Adebrelimab Combined With Famitinib and Chemotherapy in the Treatment of ES-SCLC.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanbin Zhao, MD, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-SCLC-II-018
Record Dates: First submitted 2024-02-29; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Extensive-stage Small-cell Lung Cancer
Keywords: Adebrelimab; Famitinib; Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — famitinib; Drug Therapy; Cisplatin; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuno-cherapy for extensive small cell lung cancer (Experimental): Adebrelimab in combination with famitinib and chemotherapy
  Interventions: Drug: adebrelimab; Drug: famitinib; Drug: chemotherapy

INTERVENTIONS:
Drug: adebrelimab — adebrelimab IV
  Other Names: SHR-1316
Drug: famitinib — famitinib PO
  Other Names: SHR1020
Drug: chemotherapy — chemotherapy IV
  Other Names: cisplatin/carboplatin and etoposide

SUMMARY:
This is a single arm, multi-center, phase II trial to evaluate the efficacy, and safety of adebrelimab combined with famitinib and chemotherapy for the treatment of first-line extensive stage small cell lung cancer.

DETAILED DESCRIPTION:
This study plans to recruit 40 patients with extensive-stage small cell lung disease who have not received treatment, observe and evaluate the effectiveness and safety of adebrelimab combined with famitinib and chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-80 years old, male or female
2. Patients with pathologically confirmed extensive stage small cell lung cancer (according to the Veterans Administration Lung Study Group, VALG staging)
3. Never received prior systemic therapy for extensive stage small cell lung cancer
4. Have a measurable tumour target lesion (meeting RECIST 1.1 criteria)
5. Expected survival > 3 months
6. ECOG PS: 0-1 points
7. Normal function of major organs
8. Women of childbearing potential must undergo a negative pregnancy test (βHCG) prior to initiation of treatment, and women of childbearing potential and men (who are sexually active with women of childbearing potential) must agree to use effective contraception uninterruptedly for the duration of the treatment period and for 6 months after the administration of the last therapeutic dose
9. Patients voluntarily enrolled in this study by signing an informed consent form

Exclusion Criteria:

1. Previous or concurrent other malignant tumours within 5 years, except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, superficial or non-invasive bladder cancer
2. Active tuberculosis infection, or a history of previous tuberculosis infection
3. Uncontrolled, symptomatic brain metastases that are not effectively controlled or a history of psychiatric illness that cannot be easily controlled or severe intellectual or cognitive dysfunction
4. Subjects with active, known or suspected autoimmune disease, hypothyroidism requiring only hormone replacement therapy, skin disorders not requiring systemic therapy (e.g., vitiligo, psoriasis, or alopecia areata) may be eligible for enrolment
5. Uncontrollable pleural effusion, pericardial effusion or ascites requiring repeated drainage
6. Subjects with the presence of any severe and/or uncontrolled disease
7. Imaging showing tumour invasion of large vessels or poor demarcation from large vessels
8. Susceptibility to bleeding, risk of hemoptysis, and history of significant coagulation disorders
9. History of psychotropic substance abuse, alcoholism or drug addiction
10. Active hepatitis (Hepatitis B reference: HBsAg positive with HBV DNA test value exceeding the upper limit of normal value Hepatitis C reference HCV antibody positive with HCV viral titre test value exceeding the upper limit of normal value)
11. Human immunodeficiency virus (HIV, HIV 1/2 antibody) positive
12. Patients who are unable to comply with the trial protocol or who are unable to cooperate with follow-up visits
13. Patients who, in the opinion of the investigator, should not be enrolled in the trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | up to 6 months
  Proportion of disease progression or death from randomization to 6 months of treatment.

SECONDARY OUTCOMES:
12-month progression-free survival | up to 12 months
  Proportion of disease progression or death from randomization to 12 months of treatment.
Objective Response Rate | up to 24 months
  Determined using RECIST v1.1 criteria, defined as best overall response (CR or PR) across all assessment time points during the period from enrolment to termination of trial treatment.
Disease control rate | up to 24 months
  Disease Control Rate, determined using RECIST v1.1 criteria.
Overall Survival | up to 24 months
  Defined as the time from randomization to death from any cause.
AEs | up to 24 months
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
QoL | up to 24 months
  Defined as time from randomization to deterioration on each of the EORTC QLQ-C30 symptom subscales
Progression-Free-Survival | up to 24 months
  Defined as the time from randomization to the first occurrence of disease progression with use of RECIST v1.1 or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Yanbin Zhao, MD, Principal Investigator — Harbin Medical University Cancer Hosptital

IPD SHARING:
Plan to Share IPD: No